CLINICAL TRIAL: NCT00621114
Title: Ex Vivo Microbiological Assessment of an Anti-biofilm Catheter in Acute Dialysis Application
Acronym: ABBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Dialysatoren GmbH (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Study No 2007_MBR_003; ISRCTN39140035 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2008-01-31; First posted 2008-02-22 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Hemodialysis
Keywords: Dialysis, Extracorporeal; Dialysis, Renal; Extracorporeal Dialysis; Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients in group 1 will be provided with a commercially available and CE certified standard double lumen catheter without surface coating (GamCath® catheter, No. CE 76891).
  Interventions: Device: GamCath® central venous catheter
- 2 (Experimental): Patients in group 2 will be treated with a CE certified double lumen catheter with a new antibacterial bismuth-containing surface coating (GamCath Dolphin® Protect, No. CE 90671).
  Interventions: Device: GamCath Dolphin® Protect central venous catheter

INTERVENTIONS:
Device: GamCath® central venous catheter — Choice of central venous catheter type
  Other Names: GamCath® catheter
  Arms: 1
Device: GamCath Dolphin® Protect central venous catheter — Choice of central venous catheter type
  Other Names: GamCath Dolphin® Protect
  Arms: 2

SUMMARY:
The clinical study aims at providing data on antimicrobial efficiency and a supposed additional preventive effect on catheter-related infections of a catheter with antibacterial surface coating in comparison to standard catheters without coating.

DETAILED DESCRIPTION:
Central venous catheters are increasingly used to provide long-term venous access, e.g. after failure of the primary arteriovenous fistula, and they are the first choice in case of an acute need for extracorporeal therapy. Microbial adhesions and biofilm formation have been implicated in serious infections associated with the use of indwelling catheters.

In view of the necessity to reduce catheter-related bloodstream infections and of the inadequacy of currently available antimicrobially coated devices, a new antimicrobial catheter surface was developed.

The clinical study described below aims at providing further data on antimicrobial efficiency and a supposed additional preventive effect on catheter-related infections.

ELIGIBILITY:
Inclusion Criteria:

* central venous catheter placement
* Need for extracorporeal renal replacement therapy (acute and chronic renal failure)
* Anticipated duration of dialysis therapy less than or equal to 30 days
* Age between 18 and 85 years
* Written informed consent

Exclusion Criteria:

* Known Hepatitis B Virus (HBV)/Hepatitis C Virus (HCV)/Human Immunodeficiency Virus (HIV) infection
* Known pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Bacterial colonisation of the catheter surface | after explantation

SECONDARY OUTCOMES:
venous and arterial pressure | during dialysis
catheter dwell time | at explantation
exit site appearance | at routine catheter care
blood parameters | during dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Teut Risler, Prof. Dr., Principal Investigator — Universitaetsklinikum Tuebingen
Locations (1):
- Universitaetsklinikum Tuebingen, Tübingen, Germany